CLINICAL TRIAL: NCT05563181
Title: Evaluation of a Beverage Media Campaign and Added-sugar Warning Labels Among Latinx Adults
Brief Title: Evaluation of a Beverage Media Campaign and Added-sugar Warning Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Jennifer Falbe, Associate Professor, University of California, Davis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1841319
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Attitude; Intention
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control bar code (Placebo Comparator): Viewing beverages that contain control labels (i.e., bar codes) on sugar-sweetened beverages
  Interventions: Behavioral: Control bar code label
- Warning label (Experimental): Viewing beverages that contain an added-sugar warning label (icon-plus-text yellow label that says, "WARNING: High in added sugar," on sugar-sweetened beverages
  Interventions: Behavioral: Warning label
- Control bar code + informational campaign about warning labels (Experimental): Viewing an informational campaign about warning labels followed by viewing beverages that contain control labels (i.e., bar codes) on sugar-sweetened beverages
  Interventions: Behavioral: Control bar code label; Behavioral: Informational campaign poster about added-sugar warning labels
- Warning label + informational campaign about warning labels (Experimental): Viewing an informational campaign about warning labels followed by viewing beverages that contain an added-sugar warning label (icon-plus-text yellow label that says, "WARNING: High in added sugar," on sugar-sweetened beverages
  Interventions: Behavioral: Warning label; Behavioral: Informational campaign poster about added-sugar warning labels

INTERVENTIONS:
Behavioral: Control bar code label — Viewing beverages that contain control labels (i.e., bar codes) on sugar-sweetened beverages
  Arms: Control bar code; Control bar code + informational campaign about warning labels
Behavioral: Warning label — Viewing beverages that contain an added-sugar warning label (icon-plus-text yellow label that says, "WARNING: High in added sugar," on sugar-sweetened beverages
  Arms: Warning label; Warning label + informational campaign about warning labels
Behavioral: Informational campaign poster about added-sugar warning labels — Viewing an informational campaign about added-sugar warning labels. The poster will be shown in Spanish (instead of English) if the participant reports speaking and reading in Spanish better than English.
  Arms: Control bar code + informational campaign about warning labels; Warning label + informational campaign about warning labels

SUMMARY:
The primary objective of this study is to examine differences in intentions (measured by hypothetical beverage selection) between the following conditions: (1) Control condition: Viewing beverages with a barcode, (2) viewing beverages that have an icon-plus-text warning label, "WARNING: High in added sugar", (3) viewing a campaign message about warning labels in one's preferred language + viewing beverages with a barcode, and (4) viewing a campaign message about warning labels in one's preferred language + viewing beverages with the warning label above. An additional objective is to compare other message reactions and perceptions and perceptions of SSBs (sugar-sweetened beverages) between the conditions. This study will use an online randomized controlled trial among Latino/a/x adults to assign participants to one of the above conditions.

DETAILED DESCRIPTION:
The primary objective of this study is to examine differences in intentions (measured by hypothetical beverage selection) between the following conditions: (1) Control condition: Viewing beverages with a barcode, (2) viewing beverages that have an icon-plus-text warning label, "WARNING: High in added sugar", (3) viewing a campaign message about warning labels in one's preferred language + viewing beverages with a barcode, and (4) viewing a campaign message about warning labels in one's preferred language + viewing beverages with the warning label above. An additional objective is to compare other message reactions and perceptions and perceptions of SSBs (sugar-sweetened beverages) between the conditions. This study will use an online randomized controlled trial among Latino/a/x adults to assign participants to one of the above conditions. Although this study uses prospective assignment, it is not a clinical trial because the outcomes are intentions, attitudes, and other reactions and perceptions and not behavioral or health outcomes.

Participants can take the survey in English or Spanish, but the warning labels on the beverages will always be in English. In the campaign conditions, if the participant generally speaks and reads in Spanish better than English, they will be shown the campaign message in Spanish, and otherwise, they will be shown the campaign message in English.

Within the campaign conditions, participants will be randomized to view 1 of 3 campaign posters that have different messages. Also, at the end of the questionnaire, all participants will be shown 1 of the 3 campaign message posters and asked to provide ratings of perceived discouragement (one of the 3 PME questions), how much the poster grabs attention, and how trustworthy the poster is. Following that item, all participants will view all 3 posters one after the other on the same page (shown in random order) and asked to select the one that discourages them the most from wanting to drink beverages high in added sugar.

1. Primary outcome: hypothetical selection of a sugar-sweetened beverage (SSB) for oneself.

   Analysis will use Poisson regression with robust standard errors, regressing dichotomous selection of an SSB on indicators for condition, which are described below:
   1. Main effects: Indicators for the warning label condition and campaign poster condition.
   2. To examine interaction effects: Indicators for warning label condition and campaign poster condition as well as a label by campaign interaction term.
2. Secondary outcomes: For binary outcomes, the analysis will entail the same modeling approach as above, and for continuous outcomes, the analysis will use linear regression models with the same indicators in the model. For outcomes about campaign posters, instead of including indicators for condition in the model, the analysis will include indicators for type of poster. For the question that asks participants to select the 1 poster (out of 3) that most discourages consumption, the analysis will use a chi-square goodness of fit test to see if the proportion of participants selecting any one poster differs significantly than what would be expected by chance. That model will include indicators for experimental condition. Within family of outcomes, the Holm-Bonferroni procedure will be used to adjust for multiple comparisons.

Exploratory analyses:

1. For the outcome of hypothetical selection of an SSB for one's child, the same modeling approach as specified for the primary outcome will be used.
2. Exploration of effect modification will be examined in separate models using interaction terms between condition and indicators for levels of the following characteristics: Participant reported speaking and reading better in Spanish than English, cut-points on the Short Acculturation Scale for Hispanics (SASH), household income and poverty level, gender, and educational attainment.

ELIGIBILITY:
Inclusion Criteria:

* Identifying as Latino/a/x
* Residing within the United States and U.S. territories
* Age 18+

Two panel companies will be used to recruit participants. To maximize recruitment of participants who prefer Spanish over English, through one of the panel companies, eligibility will be restricted to participants reporting that Spanish was their first language and through the second panel, a quota will be used to aim for ≥50% who prefer Spanish over English. For the second panel, additional quotas will be used to maximize gender balance and inclusion of parents: ≤60 percent women, and ≥50% with a child age 2-17. Quotas may need to be adjusted to obtain desired sample size.

Exclusion Criteria for main analysis:

* Failing attention check question
* Speeding (finishing survey in <33% of the median completion time)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2275 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Intention to purchase a sugar-sweetened beverage in a hypothetical selection task (not a scale) | Approximately 0.5-2 minutes
  Measured in a hypothetical beverage selection task in which participants are shown supermarket shelves containing a variety of sugar-sweetened and non-sugar-sweetened beverages, labeled according to condition. Participants will be asked to select the one beverage they would want to purchase for themselves, and this outcome will be dichotomized as hypothetical selection of an SSB or not. Adapted from doi: 10.2105/AJPH.2021.306488.

SECONDARY OUTCOMES:
Intention to consume sugar-sweetened beverages and water in the next 4 weeks (there is no scale title) | ≤20 minutes
  Assessed via questionnaire items asking likelihood of consumption (5-point scale: 1=not at all to 5=extremely likely). Adapted from doi: 10.2105/AJPH.2021.306488.
Scale title: University of North Carolina (UNC) Perceived message effectiveness (PME) | ≤20 minutes
  Adapted 3-item UNC PME scale (each item--concern, unpleasant, and discourage--has a 5-point scale from strongly disagree=1 to strongly agree=5, and all item scores are averaged for the overall PME score [the higher the score, the higher the perceived effectiveness].) Adapted from doi: 10.1093/abm/kay080.
Noticing the label (not a scale) | ≤20 minutes
  Questionnaire item adapted from doi: 10.1016/j.ypmed.2022.107090. Response options are yes (indicating noticing), no, and I don't know. If yes is selected, categories of topics are presented from which the participant can select. Only one option is the correct option (indicating noticing).
Outcome expectations re: sugar-sweetened beverages increasing risk of type 2 diabetes, heart disease, and tooth decay (there is no scale title) | ≤20 minutes
  Questionnaire items (5-point scale from 1=strongly disagree to 5=strongly agree) adapted from doi: 10.1016/j.ypmed.2022.107090
Perception of learning something new from the label (not a scale) | ≤20 minutes
  Questionnaire item (dichotomous yes/no response) adapted from doi: 10.1016/j.ypmed.2022.107090
Anticipated social interaction about the label (there is no scale title) | ≤20 minutes
  Questionnaire item (5-point scale from 1=not at all likely to 5=extremely likely) adapted from doi: 10.3390/ijerph121013195
Support for policy requiring labels (there is no scale title) | ≤20 minutes
  Questionnaire item (5-point scale from 1=strongly oppose to 5=strongly support) adapted from doi: 10.1016/j.ypmed.2022.107090
Reactions to poster: Perception that informational campaign poster discourages consumption of beverages high in added sugar (adapted item from the UNC PME Scale), grabs attention (no scale title), and is trustworthy (no scale title) | ≤20 minutes
  Questionnaire items (discourage: 5-point scale from 1=strongly disagree to 5=strongly agree and attention and trustworthy: 5-point scale from 1=not at all to 5=a great deal) adapted from doi: 10.1016/j.ypmed.2022.107090
Selection of informational campaign that most discourages consumption of beverages high in added sugar (not an scale) | ≤20 minutes
  Questionnaire item (categorical responses) adapted from doi: 10.1016/j.ypmed.2022.107090

OTHER OUTCOMES:
Intention to purchase a sugar-sweetened beverage for one's child under the age of 18 in a hypothetical selection task (not a scale) | Approximately 0.5-2 minutes
  Measured in a hypothetical beverage selection task in which participants are shown supermarket shelves containing a variety of sugar-sweetened and non-sugar-sweetened beverages, labeled according to condition. Participants will be asked to select the one beverage they would want to purchase for their child, and this outcome will be dichotomized as hypothetical selection of an SSB or not. Adapted from doi: 10.2105/AJPH.2021.306488.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Falbe, Principal Investigator — UC Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolf EC, Hall MG, Schillinger D, Krieger J, Woo Baidal JA, Solar S, Lin C, Falbe J. Online RCT of Added-Sugar Warning Labels and Spanish-English Label Education. Am J Prev Med. 2025 Oct;69(4):107966. doi: 10.1016/j.amepre.2025.107966. Epub 2025 Jul 4. PMID 40617305